CLINICAL TRIAL: NCT04121494
Title: A Phase I Clinical Trial to Compare the Safety and Immunogenicity of Candidate TB Vaccine ChAdOx1 85A Administered by the Aerosol Inhaled Route and the Intramuscular Route in Healthy Adult Subjects
Brief Title: ChAdOx1 85A Aerosol Versus Intramuscular Vaccination in Healthy Adults (TB039)
Acronym: TB039
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: François Spertini (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor-Investigator, François Spertini, médecin-chef, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHADOX
Record Dates: First submitted 2019-08-20; First posted 2019-10-10 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Mycobacterium Tuberculosis, Protection Against; Tuberculosis
Keywords: ChAdOx1 85A; Tuberculosis; vaccination; BCG; Mucosal; Inhaled vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: Stage I - dose escalation study (Arms A,B,C) Stage II - experimental arms: randomized (Arms D,E), parallel (Arm F)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking for Arms D,E Non-masking for Arms A,B,C,F
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): BCG-vaccinated, 1x10^9 vp, aerosol
  Interventions: Biological: ChadOx1 85A - aerosol
- Group B (Experimental): BCG-vaccinated, 5x10^9 vp, aerosol
  Interventions: Biological: ChadOx1 85A - aerosol
- Group C (Experimental): BCG-vaccinated, 1x10^10 vp, aerosol
  Interventions: Biological: ChadOx1 85A - aerosol
- Group D (Experimental): BCG-vaccinated, highest tolerated dose aerosol + placebo IM; Randomized with Group E, blind
  Interventions: Biological: ChadOx1 85A - aerosol
- Group E (Experimental): BCG-vaccinated, highest tolerated dose IM + placebo aerosol; Randomized with Group D, blind
  Interventions: Biological: ChadOx1 85A - IM
- Group F (Experimental): BCG-non vaccinated, highest tolerated dose, aerosol
  Interventions: Biological: ChadOx1 85A - aerosol

INTERVENTIONS:
Biological: ChadOx1 85A - aerosol — Aerosol administration through the Omron MicroAIR NE-U22 nebuliser
  Arms: Group A; Group B; Group C; Group D; Group F
Biological: ChadOx1 85A - IM — Intramuscular administration
  Arms: Group E

SUMMARY:
This is a dose escalating and a paired-placebo design study to describe the safety and immunogenicity profile of candidate TB vaccine ChAdOx1 85A given by aerosol inhaled vaccination versus intramuscular (IM) vaccination in adult healthy volunteers.

It is postulated that the aerosol inhaled route is practical and feasible and has an acceptable safety profile, comparable to the systemic safety profile of the IM route of administration of ChAdOx1 85A in adult healthy volunteers, and that the aerosol inhaled route of administration will induce greater mucosal immunity and comparable systemic immunity when compared to the IM (systemic) route of administration in these volunteers.

Volunteers are followed on a regular basis for safety and immunogenicity, with blood analysis for biological safety tests and immune tests.

DETAILED DESCRIPTION:
Background:

Mycobacterium tuberculosis (M.tb) is a pathogen with worldwide preponderance which infects humans and causes tuberculosis (TB), a transmissible disease resulting in very high mortality and morbidity. A third of the world's population is latently infected with M.tb, and these people carry a 10% lifetime risk of developing active life-threatening disease. In 2015, there were 10.4 million new cases worldwide and 1.8 million people died of TB. Co-infection with human immunodeficiency virus (HIV) greatly increases risk of TB reactivation and death. Diagnosis is challenging and drug treatment can be prolonged, harmful, costly and complex. For these reasons an effective TB vaccine is a global public health priority.

The Bacille Calmette-Guérin (BCG) vaccine is the only licensed TB vaccine and it has been administered globally to several billion people over a 90 year period. Although it does not protect against pulmonary TB in endemic areas, it is effective in preventing disseminated TB disease including tuberculous meningitis in childhood. Recently, heterologous "prime-boost" vaccination strategies, in which two different candidate vaccines expressing antigens in common are given weeks or months apart, have generated strong and sustained cellular immune responses correlating with an M.tb protective effect in preclinical animal models. In such a "prime-boost" strategy, BCG would therefore be an ideal priming vaccine.

ChAdOx1 85A is a new adenoviral vaccine based on a vector that is a chimpanzee adenovirus isolate Y25 expressing the M.tb antigen 85A. Adenoviruses are attractive candidates for use as viral vectors and have been used as vaccine vectors for a number of conditions; however the use has been limited by the high level of anti-vector immunity present in humans in whom adenovirus is a ubiquitous infection. This has led to the consideration of simian adenoviruses, which are not known to cause pathology or illness in humans and to which the prevalence of anti-vector antibodies is low.

The route of M.tb infection is by inhalation of aerosolised infectious droplets containing tubercle bacilli, leading to the establishment of primary infection in the lung, which has a distinct mucosal immune system characterized by bronchus associated lymphoid tissue (BALT), which is well adapted to encounter and process such antigens. Immunising via the airway should therefore have the advantage, over other routes, of eliciting protective immune responses in the lung mucosa. There is data from preclinical animal models with virally vectored vaccines to suggest that immunising the respiratory mucosa may give superior protection against respiratory diseases. The inhaled route is a well-established route of drug delivery for humans and there are numerous perceived advantages of aerosol inhaled vaccination.

This trial will be the first to evaluate the safety and immunogenicity of candidate TB vaccine ChAdOx1 85A given by aerosol inhaled vaccination. Using a paired-placebo design, the trial will investigate aerosol vaccination compared to intramuscular vaccination, the latter for which initial safety data has already been collected and from which the dosing regimen for this trial has been chosen.

Objective:

The study aims to describe the safety and immunogenicity profile for ChAdOx1 85A given by aerosol inhaled vaccination versus intramuscular (IM) vaccination in adult healthy volunteers.

Methods:

Thirty-nine subjects will be enrolled into the trial: 29 BCG-vaccinated and 10 BCG-naïve.

Nine BCG-vaccinated healthy volunteers will receive the ChAdOx1 85A vaccine by aerosol inhaled vaccination at three different dose levels (3 volunteers per dose levels, Groups A-B-C). Based on the safety profile and immunogenicity results obtained in Groups A, B and C, the highest tolerated dose will be determined, and a decision made as to which dose to use for subsequent Groups.

The next 20 BCG-vaccinated subjects will be blinded and randomised in Groups D and E: volunteers randomised to the intervention group (D, inhaled aerosol) will receive a concurrent intramuscular saline injection, while volunteers in the control group (E, intramuscular) will receive a concurrent dose of inhaled saline. This design has the added benefit of allowing a distinction to be made between any adverse events attributable to the method (including nebuliser device) of vaccine delivery and those attributable to the inhaled investigational medicinal product itself.

In parallel to enrolment of Groups D and E, 10 BCG naïve subjects will be enrolled in Group F to receive the highest tolerated dose by aerosol inhaled vaccination.

After vaccination (day 0), volunteers will then follow a schedule of visits over the six months (day 1, day 7, day 14, day 28, day 84 and day 168), for safety and immunological follow-up via blood tests and physical examination. Moreover, at day 14, volunteers will undergo a bronchoscopy to check for signs of inflammation or other damage and to obtain a bronchoalveolar lavage sample and lymph node cytopunction.

Impact:

The overall investigational approach with ChAdOx1 85A trials is to develop an effective prime-boost vaccination strategy to prevent TB infection, with BCG as the priming vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-55 years.
* Give informed consent as documented by signature.
* Screening Interferon-Gamma release assay (IGRA) negative.
* Chest radiograph normal.
* Prior vaccination with BCG (except Group F).
* No relevant findings in medical history or on physical examination.
* Allow the Investigators to discuss the individual's medical history with their GP, if appropriate.
* Use effective double contraception for the duration of the trial period (females and males).
* Refrain from blood donation during the trial.
* Able and willing (in the Investigator's opinion) to comply with all the trial requirements.

Exclusion Criteria:

* Previously resident for more than 12 consecutive months in a highly endemic area (tropical) where significant TB and non-tuberculous mycobacterial exposure is likely.
* Participation in another research trial involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the trial period.
* Participation in a clinical trial involving vaccination with an adenovirus vector (such as Ebola or HIV trials)
* Prior vaccination with any candidate TB vaccine.
* Vaccination with any live, attenuated vaccine within 28 days prior to enrolment.
* Vaccination with any subunit or killed vaccine within 14 days prior to enrolment (influenza vaccination is encouraged prior to participation).
* Prior vaccination with BCG (Group F only).
* Administration of immunoglobulins and/or any blood products within the three months preceding the enrolment.
* Clinically significant history of skin disorder, allergy, atopy, immunodeficiency (including HIV), cancer (except basal cell carcinoma or carcinoma in situ), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse.
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents.
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial agent, sedative drugs, or any local or general anaesthetic agents.
* Pregnancy, lactation or intention to become pregnant during trial period.
* Any respiratory disease, including perennial asthma, non-controlled seasonal allergic asthma
* Smoking more than 3 cigarettes/day.
* Clinically significant abnormality on screening chest radiograph.
* Clinically significant abnormality of spirometry.
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy.
* Current use of any medication taken through the inhaled route.
* Clinical, radiological, or laboratory evidence of current active TB disease.
* Past treatment for TB disease.
* Any clinically significant abnormality of screening blood or urine tests.
* Positive HBsAg, HCV or HIV antibodies.
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the trial or impair interpretation of the trial data.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Safety - (serious) adverse events | Day 0 to Day 168
  Frequency, incidence and nature of Adverse Events (AE) and Serious Adverse Events (SAE)

SECONDARY OUTCOMES:
Immunogenicity | Day 0 to 168
  Characterization of cell mediated and humoral immune markers in response to vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
availability of study protocol
Supporting Information: Study Protocol
Time Frame: immediately without limit in time

REFERENCES:
- [Derived] Crisan-Dabija R, Grigorescu C, Pavel CA, Artene B, Popa IV, Cernomaz A, Burlacu A. Tuberculosis and COVID-19: Lessons from the Past Viral Outbreaks and Possible Future Outcomes. Can Respir J. 2020 Sep 5;2020:1401053. doi: 10.1155/2020/1401053. eCollection 2020. PMID 32934758